CLINICAL TRIAL: NCT06183684
Title: Early Feasibility Study (EFS) Laplace Transcatheter Tricuspid Valve Replacement (TTVR) System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laplace Interventional, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLN-002
Record Dates: First submitted 2023-12-07; First posted 2023-12-27 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Tricuspid Valve Replacement (Experimental): Transcatheter replacement of the native tricuspid valve with the Laplace bioprosthesis
  Interventions: Device: Laplace TTVR System

INTERVENTIONS:
Device: Laplace TTVR System — Transcatheter Tricuspid Valve Replacement (TTVR) System for the treatment of severe, symptomatic tricuspid regurgitation

SUMMARY:
The objective of the study is to assess the safety and technical feasibility of the Laplace Transcatheter Tricuspid Valve Replacement (TTVR) System

DETAILED DESCRIPTION:
Early Feasibility (EFS), prospective, single-arm, multi-center study to evaluate safety and technical feasibility of the Laplace TTVR System in the treatment of severe, symptomatic tricuspid regurgitation patients.

ELIGIBILITY:
Inclusion Criteria:

1. 22 - 90 years of age at the time of the study procedure
2. Symptomatic tricuspid regurgitation despite being adequately treated with optimal medical therapy by the Local Heart Team for at least 30 days prior to the time of study consent.
3. Severe, massive or torrential tricuspid regurgitation determined by qualifying transthoracic echocardiogram (TTE) and/or transesophageal echocardiogram (TEE) using the 5-grade classification.
4. Candidate felt suitable for transcatheter tricuspid valve replacement as determined by the local heart team and confirmed by the patient selection committee. For patients with pre-existing trans-tricuspid pacemaker or ICD leads, the local heart team shall include an electrophysiologist.
5. Subject or legally authorized representative has provided informed consent and agrees to return for all required post-procedure follow-up visits

Exclusion Criteria:

1. Estimated life expectancy of less than 12 months
2. PVR >5 Wood units
3. Echocardiographic evidence of severe right ventricular dysfunction
4. Severe aortic, mitral and/or pulmonic valve stenosis and/or regurgitation requiring treatment
5. Presence of significant congenital heart disease including but not limited to hemodynamically significant atrial septal defect, RV dysplasia, and arrhythmogenic RV.
6. Any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery, within last 30 days. Implant or revision of any rhythm management device (CRT or CRT-D) or implantable cardioverter-defibrillator or leadless pacemaker within 90 days prior to the study procedure
7. Stroke or other major cerebrovascular event within 90-days prior to index procedure
8. Untreated clinically significant coronary artery disease requiring revascularization, recent (within last 30 days) acute coronary syndrome or myocardial infarction.
9. Bleeding disorders including thrombocytopenia or platelet count <70,000 mm3 or thrombocytosis (platelet count >700,000 /mm3)
10. Current or planned pregnancy within next 12 months for women of childbearing potential
11. Active or recent endocarditis within last 90 days or, sepsis/ other systemic infection requiring oral or intravenous antibiotics within last 30 days
12. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements. Any patient considered to be vulnerable.
13. Left ventricular ejection fraction (LVEF) < 30%

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Technical success | During procedure
  Successful valve implantation

SECONDARY OUTCOMES:
Procedural success | During procedure
  Tricuspid regurgitation of moderate or less
Device success | 30-days post-procedure
  Freedom from reintervention due to device related complications

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Tucson Medical Center, Tucson, Arizona
  - Kaiser Permanente, San Francisco, California
  - Piedmont Hospital, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Providence Heart Institute, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No